CLINICAL TRIAL: NCT03389191
Title: A Clinical Trial of Oral Acyclovir in Viral Uveitis
Brief Title: A Clinical Trial of Acyclovir for Viral Uveitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiaomin Zhang (Other)
Responsible Party: Sponsor-Investigator, Xiaomin Zhang, MD, PhD, Principal Investigator, Clinical Professor, Tianjin Medical University
Organization: Tianjin Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017KY-07
Record Dates: First submitted 2017-12-27; First posted 2018-01-03 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-04

CONDITIONS: Uveitis
MeSH Terms: conditions — Uveitis | interventions — Acyclovir

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | US Export: No

ARMS (1):
- Patients with Viral Uveitis (Experimental): Oral acyclovir 100 mg three times a day (TID).
  Interventions: Drug: Acyclovir

INTERVENTIONS:
Drug: Acyclovir

SUMMARY:
This project is designed to test the hypothesis that acyclovir is clinically useful for patients with refractory viral uveitis.

DETAILED DESCRIPTION:
Approval of the study was obtained from the hospital's ethical committee. The study design and methodology followed the tenets of Declaration of Helsinki. All patients were provided with written informed consent and received a thorough explanation of the study design, aims, benefits and potential risks. This is a prospective non-comparative interventional study.

Aqueous humor samples were collected from participants to virus detection. Participants will take oral acyclovir 100 mg three times a day and data will be collected prospectively with regard to ophthalmologic outcomes. Study participants will be followed for up to 12 months to determine efficacy, and an additional 30 days for safety reports. Descriptive statistics will be gathered on participant demographics, uveitis characteristics, change in immunosuppressive medications, number of responders, ophthalmologic measures and change in corticosteroid dose during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and above.
* Chronic, vision threatening viral uveitis.
* Patients can't tolerate hormone therapy bacause of drug side effects.
* Consent to undergo anterior chamber tap and give aqueous for the study.
* Able to undergo relevant tests.
* Able to come for subsequent follow-up visits.
* Ability to provide informed consent.

Exclusion Criteria:

* Patients who are allergic to ayclovir.
* Immunocompromised patients
* Positive for HIV, Hep B and Hep C
* Not keen on participating in the study
* Patients who are incapable, either by law or mental state, of giving consents in their own right.
* Patients who are either unable or unwilling to keep scheduled appointments and adhere to the other aspects of the protocol.
* Patients who are pregnant or breastfeeding.
* Any other specified reason as determined by the clinical investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Mean and median change in best corrected visual acuity in logMAR | 12 weeks
  Mean and median change in best corrected visual acuity in logMAR

SECONDARY OUTCOMES:
Number of participants who experience a recurrence | 12 weeks
  Number of participants who experience a recurrence
Length of time to quiescence | 12 weeks
  Length of time to quiescence
Ability to taper concomitant immunosuppressive medications | 12 weeks
  Ability to taper concomitant immunosuppressive medications
Number and severity of systemic and ocular toxicities and adverse events | 12 weeks
  Number and severity of systemic and ocular toxicities and adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Xiaomin Zhang, M.D., Study Director — Tianjin Medical University Eye Hospital
Locations (1):
- Tianjin Medical University Eye Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The study protocol,statistical analysis plan,informed consent form and clinical study report are to be shared with other researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will become available starting 6 months after publication.
Access Criteria: Study protocol, statistical analysis plan and informed Consent form can be shared with other researchers. And researchers will review requests and criteria for reviewing requests.